CLINICAL TRIAL: NCT02564419
Title: Early Feasibility Study of a Medtronic Activa PC+S System for Persons Living With Spinal Cord Injury
Brief Title: Brain Machine Interface (BMI) in Subjects Living With Quadriplegia
Acronym: BMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Jagid (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Jonathan Jagid, Associate Professor of Neurological Surgery, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20150244
Record Dates: First submitted 2015-08-18; First posted 2015-09-30 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Medtronic Activa PC + S is a multi-programmable primary cell neurostimulator that records bioelectric data and deliver electrical stimulation through leads implanted in the brain.
Masking Description: Participants will be undergoing a unilateral implantation of the Medtronic Active PC+S with unilateral subdural strip electrodes over the motor cortex. They will receive 24 sessions over a 3-6 month period which consists of external stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Medtronic Activa PC+S (Experimental): Objective of this pilot phase early feasibility study is to assess the safety and feasibility of Medtronic Activa PC+S implant (device) by;
  1. Evaluating the ability of the Activa PC+S system to sense ECoG signals in subjects living with quadriplegia (C5 or C6 level).
  2. Assessing the feasibility of activating fundamental upper extremity muscles to reproduce hand grasp.
  These are important first steps towards creating and designing a device that can enhance or assist in performing activities of daily living (ADL) in the life of these subjects. Attachment 15.3
  Interventions: Device: Medtronic Activa PC+S

INTERVENTIONS:
Device: Medtronic Activa PC+S — Upon consent, the good candidates will undergo surgical screening that includes a full neurological workup and baseline functional assessment. Subjects that demonstrate feasibility for control will undergo surgery for unilateral implantation of the Activa PC+S as well as the implantation of unilateral subdural strip electrodes (Resume II, model 3587A) over the motor cortex. After 24 hour observation in the hospital, subjects will participate in 24 distinct sessions or visits of testing over a 3-6 month period. During these visits, the sensing, decoding of the implanted device (Activa PC+S) as well as the external stimulation components (Bioness H200) and parameters will be tested and benchmarked. Subjects will participate for 24 sessions and continue to participate in the study until the end of life of the device, at which point the subject may elect to undergo an explant at that time.

SUMMARY:
In this study, investigators will show proof-of-concept that brain signals can be used in real-time, closed-loop mode to trigger stimulation for hand function. Subjects will undergo surgery to implant a unilateral subdural strip electrode (Resume II, Model 3587A) over the motor cortex. These electrodes implanted in the brain will enable bioelectrical data recording (sensing) from the brain to the implanted Activa PC+S. The cortical sensing data will be

1. either processed in the Activa PC+S; or
2. off-loaded via the Nexus D communication device (Medtronic) to a computer.

ELIGIBILITY:
Inclusion Criteria:

* AIS Grades A & B
* Level of Injury C5 or C6
* Local Community dwelling
* Stable chronic injury
* Stable health status and upper extremities
* Completion of Clinical Protocol 01

Exclusion Criteria:

* Coagulopathy
* Anticoagulation
* Pregnancy

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
AIS Motor Score | Up to 2 years
  American Spinal Injury Association (ASIA) Impairment Scale (AIS) Motor scores has a score totaling 0-50 for the upper limbs and 0-50 for the lower limbs with the lower score indicating greater motor impairment
AIS Sensory Score | Up to 2 years
  AIS Sensory scores has a score totaling 0-56 points for light touch and pin prick modalities for a total of a maximum of 112 points per side of the body. The lower scores indicate greater sensory impairment.
SF-36 scores | Up to 2 years
  Short Form 36 (SF-36) is a 36 item self-report health questionnaire
Muscle Force Test | Up to 2 years
  0. No movement;1.Palpable contraction, no visible movement; 2. Movement but only with gravity eliminated; 3. Movement against gravity; 4. Movement against resistance but weaker than normal; 5. Normal power
Range of Motion | Up to 2 years
  Joint Range of Motion for both active and passive for Flexion and extension
SCIM III (Spinal Cord Independence Measure) | Up to 2 years
  Self-report independence for daily activities of living scored from 1-6
JTT Hand Function Test | Up to 2 years
  Functional timed activities such as hand writing, page turning, lifting small objects, feeding, stacking checkers, lifting light cans and lifting heavy cans
Pinch Grip Strength | Up to 2 years
  Measurement of grip strength throughout training
Modified Ashworth Scale | Up to 2 years
  Muscle tone scored during stretch from 0 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Jagid, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami School of Medicine/Miami Project to Cure Paralysis, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis KC, Meschede-Krasa B, Cajigas I, Prins NW, Alver C, Gallo S, Bhatia S, Abel JH, Naeem JA, Fisher L, Raza F, Rifai WR, Morrison M, Ivan ME, Brown EN, Jagid JR, Prasad A. Design-development of an at-home modular brain-computer interface (BCI) platform in a case study of cervical spinal cord injury. J Neuroeng Rehabil. 2022 Jun 3;19(1):53. doi: 10.1186/s12984-022-01026-2. PMID 35659259